CLINICAL TRIAL: NCT00383981
Title: Lipid Peroxidation in Workers Exposed to Al,Ga,In,As,and Sb in Optoelectronic Industry
Status: Completed | Type: Observational
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Other Study IDs: KMUH-IRB-950067
Record Dates: First submitted 2006-10-03; First posted 2006-10-04 (Estimated); Last update posted 2006-10-04 (Estimated); Status verified 2006-04

CONDITIONS: Urine
Keywords: malondialdehyde optoelectronic vitamin complex

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
To investigate whether exposure to Al, Ga, In, As, and Sb induces lipid peroxidation in humans. Whole blood and urine levels of 170 workers were analysed by use of ICP-MS. MDA, the product of lipid peroxidation was determined by HPLC

DETAILED DESCRIPTION:
If MDA as an index of lipid peroxidation can be induced by these metals. We will suggest reducing exposure to these metals

ELIGIBILITY:
Inclusion Criteria:

* Optoelectronic workers

Exclusion Criteria:

* Office workers

Ages: 22 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 170
Dates: Start 2003-03; Study Completion 2003-12

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Hsiung Liao, Master, Principal Investigator — Department of Public Health Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University, Kaohsiung City, Taiwan